CLINICAL TRIAL: NCT02413840
Title: Evaluation, Psychological Intervention and Follow-up Study of Anxiety and Depression in Stable Chronic Obstructive Pulmonary Disease Patients
Brief Title: Evaluation, Psychological Intervention and Follow-up Study of Anxiety and Depression in Stable COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huimin Gong (Other)
Responsible Party: Sponsor-Investigator, Huimin Gong, Resident, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMU900314
Record Dates: First submitted 2015-02-04; First posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: COPD; Anxiety; Depression
Keywords: COPD; Baduanjin qigong; depression; anxiety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baduanjin qigong group (Experimental): Doing exercise of Baduanjin qigong under the guidance of medical staff;psychological counseling at the same time.
  Interventions: Behavioral: Baduanjin qigong
- control group (No Intervention): Psychological counseling only.

INTERVENTIONS:
Behavioral: Baduanjin qigong
  Arms: Baduanjin qigong group

SUMMARY:
This study expect to investigate psychological intervention (Baduanjin qigong) in COPD patients combined with anxiety and/or depression.

DETAILED DESCRIPTION:
Anxiety and depression is one of the most common complications of COPD patients.This research use psychological questionnaires to evaluate the stage of COPD patients with anxiety and/or depression(asymptomatic, subclinical，clinical). The subclinical type will divided into the treatment group of Baduanjin qigong，and the control group. Two groups are all receive the same psychological counseling, the treatment group also receive further treatment of Baduanjin qigong under the guidance of medical staff. The treatment along for 1 year. Two groups were followed up for 2 years, dynamically observe the stage of anxiety and depression,the number of exacerbations,lung function,etc.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of COPD
* In stable phase
* FEV1%predicted <80.

Exclusion Criteria:

* Cancer
* Severe cerebrovascular disease
* Severe arrhythmia,cardiac insufficiency
* Alzheimer's disease
* Mental illness
* Severe liver disfunction
* Severe renal disfunction
* Physical activity disable.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
stage of anxiety and depression ((Hospital Anxiety and Depression Scale) | one year
  use psychological questionnaires(Hospital Anxiety and Depression Scale,etc)to evaluate the stage of anxiety and/or depression

SECONDARY OUTCOMES:
the number of acute exacerbations | one year
lung function (pulmonary function test(20 minutes after inhaled 400ug albuterol),the forced expiratory volume in 1 second(FEV1)will be detected) | one year
  use pulmonary function test(20 minutes after inhaled 400ug albuterol),the forced expiratory volume in 1 second(FEV1)will be detected.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, Study Chair — Capital Medical University
Locations (1):
- Beijing institute of respiratory diseases, Beijing, China